CLINICAL TRIAL: NCT04582084
Title: Assessment of Treatment Safety and Quality of Life in Patients Receiving Etanercept Biosimilar for Autoimmune Arthritis (ASQA): a Multicenter Post-marketing Surveillance Study
Brief Title: Assessment of Treatment Safety and Quality of Life in Patients Receiving Etanercept Biosimilar for Autoimmune Arthritis
Acronym: ASQA
Status: Completed | Type: Observational
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Other Study IDs: ETA.ARY.AJ.93
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Etanercept; Biosimilar; Safety; Quality of life; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — Etanercept; etanercept biosimilar SB4

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune Arthritis: Patients with autoimmune arthritis, including rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis, receiving biosimilar etanercept in real-world settings
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Patients received biosimilar etanercept 25 mg twice weekly or 50 mg once weekly.
  Other Names: Biosimilar etanercept; Altebrel

SUMMARY:
In this open-label, multi-center, observational, post-marketing surveillance study, patients with ankylosing spondylitis, psoriatic arthritis, or rheumatoid arthritis received biosimilar etanercept 25 mg twice weekly or 50 mg once weekly in real-world settings. Safety and effectiveness of biosimilar etanercept were evaluated in study participants for a duration of up to 12 months.

DETAILED DESCRIPTION:
In this open-label, multi-center, observational, post-marketing surveillance study, patients with ankylosing spondylitis, psoriatic arthritis, or rheumatoid arthritis received biosimilar etanercept 25 mg twice weekly or 50 mg once weekly in real-world settings. Safety and effectiveness of biosimilar etanercept were evaluated in study participants for a duration of up to 12 months. Patient information was recorded in four notebooks, and each notebook had three sections, one section for each month. The first section of notebook I contained demographic information, pregnancy and lactation status in female patients, cigarette smoking and alcohol consumption, and past medical history. All safety and effectiveness outcomes were recorded at the appropriate sections of the notebooks.

ELIGIBILITY:
Inclusion Criteria:

* Adults with the diagnosis of rheumatoid arthritis, ankylosing spondylitis, or psoriatic arthritis receiving biosimilar etanercept (either 25 mg or 50 mg) for their medical condition.

Exclusion Criteria:

* No strict exclusion criteria were applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis, ankylosing spondylitis, or psoriatic arthritis receiving biosimilar etanercept (either 25 mg or 50 mg) for their medical condition were eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of adverse events | Throughout the study period (up to 12 months for each patient)
  All adverse events, including serious adverse events, are reported using system organ classes and preferred terms of the medical dictionary for regulatory activities (MedDRA Desktop Browser 4.0 Beta).

SECONDARY OUTCOMES:
Health assessment questionnaire (HAQ)-score | Baseline, 3, 6, 9, and 12 months
  Health assessment questionnaire (HAQ) is a functional test used in patients with a wide variety of rheumatic diseases, including rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis. HAQ score ranges from 0 to 3, with higher scores indicating more severe functional disability.
Pain score | Baseline, 3, 6, 9, and 12 months
  Pain assessment is performed on a scale of 0 to 10, with higher scores indicating greater pain.
Patient global assessments of disease activity (PGA) | 3, 6, 9, and 12 months
  Patient global assessment of disease activity (PGA) is a very common patient reported outcome measure used in rheumatic disorders. PGA assessment is performed on a scale of 0 to 10, with higher scores indicating higher disease activity.
Physician global assessment of disease activity (PhGA) | 3, 6, 9, and 12 months
  Physician global assessment of disease activity (PhGA) is used to assess disease severity by physicians. PhGA assessment is performed on a scale of 0 to 10, with higher scores indicating higher disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmadreza Jamshidi, Principal Investigator — Rheumatology Research Center, Tehran University of Medical Sciences
Locations (10):
- Iran (10):
  - Connective Diseases Research Center, Tabriz University of Medical Sciences, Tabriz, East Azerbaijan Province
  - Hafez Hospital, Shiraz, Fars
  - Razi Hospital, Rasht, Gilan Province
  - Ghaem Hospital, Mashhad, Khorasan
  - Golestan Hospital, Ahvāz, Khouzestan
  - Alzahra Hospital, Isfahan
  - Personal Office, Isfahan
  - Kerman University of Medical Sciences, Kerman
  - Personal Office, Shiraz
  - Rheumatology Research Center, Tehran University of Medical Sciences, Tehran

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified individual participant data (IPD) will be shared.
Time Frame: Starting 6 months after publication.
Access Criteria: Data would be shared upon reasonable request from the Study Principal Investigator, without any specific criteria:
  Ahmadreza Jamshidi Rheumatology Research Center, Tehran University of Medical Sciences, Tehran, Iran Email: dr.ahmadreza.jamshidi@gmail.com Tel: +982188220065

REFERENCES:
- [Derived] Gharibdoost F, Salari AH, Salesi M, Ebrahimi Chaharom F, Mottaghi P, Hosseini M, Sahebari M, Nazarinia M, Mirfeizi Z, Shakibi M, Moussavi H, Karimifar M, Mowla K, Karimzadeh H, Anjidani N, Jamshidi A. Assessment of Treatment Safety and Quality of Life in Patients Receiving Etanercept Biosimilar for Autoimmune Arthritis (ASQA): A Multicenter Post-marketing Surveillance Study. Adv Ther. 2021 Feb;38(2):1290-1300. doi: 10.1007/s12325-020-01611-8. Epub 2021 Jan 11. PMID 33432540